CLINICAL TRIAL: NCT00921791
Title: Efficacy of Home Blood Pressure Monitoring to Improve Blood Pressure Control: a Randomized Controlled Trial With Ambulatory Blood Pressure Measurement
Brief Title: Efficacy of Home Blood Pressure Monitoring (MONITOR Study)
Acronym: MONITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sandra Costa Fuchs, MD, PhD, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: GPPG 04465
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Home Blood Pressure Monitoring; Ambulatory Blood Pressure Monitoring; Pharmaceutical care
MeSH Terms: conditions — Hypertension | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Home Blood Pressure Monitoring (Experimental): Automatic oscillometric device for blood pressure measurement at home plus usual care.
  Interventions: Device: HBPM
- HBPM and Pharmaceutical care (Experimental): Automatic oscillometric device for blood pressure measurement at home and consultations with the pharmacists plus usual care.
  Interventions: Device: HBPM and Pharmaceutical care
- Pharmaceutical care (Active Comparator): Consultations with the pharmacists plus usual care.
  Interventions: Behavioral: Pharmaceutical care
- Control (Active Comparator): Usual care: participants are instructed to keep on their current antihypertensive medication and receive non-pharmacological recommendations for hypertension treatment.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: HBPM — Automatic oscillometric device for home blood pressure measurement and usual care.
  Arms: Home Blood Pressure Monitoring
Device: HBPM and Pharmaceutical care — Automatic oscillometric device for blood pressure measurement at home and consultations with the pharmacists
  Other Names: HBPM
  Arms: HBPM and Pharmaceutical care
Behavioral: Pharmaceutical care — consultations with the pharmacists
  Other Names: DADER method
  Arms: Pharmaceutical care
Other: Usual care — Consultation with the physician.
  Other Names: Usual clinical practice.
  Arms: Control

SUMMARY:
High blood pressure is the main risk factor for cardiovascular disease worldwide,but its control rate is unsatisfactory. Home Blood Pressure Monitoring (HBPM) with automatic oscillometric devices and pharmaceutical care have been proposed as interventions to increase therapeutic compliance and to guide treatment decisions.

The purpose of this study is to evaluate the effect of HBPM and of pharmaceutical care in blood pressure control measured through 24h ambulatory blood pressure monitoring (ABPM).

DETAILED DESCRIPTION:
Home Blood Pressure Monitoring (HBPM) and Pharmaceutical care have been proposed to improve therapeutic compliance and to guide treatment decisions, but their effects on BP control are still under debate.

This is a factorial randomized controlled trial including adult hypertensive patients under drug treatment but with office BP and 24h ABPM uncontrolled. Participants will be allocated to one of four groups: HBPM; HBPM and Pharmaceutical care; Pharmaceutical care; or control. All participants will receive usual care for high blood pressure. Participants will be followed for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Office BP ≥140/90 mm Hg
* 24h ABPM hypertension BP ≥130/80 mm Hg
* using at least one antihypertensive drug

Exclusion Criteria:

* BP ≥ 180 / 110 mmHg)
* major cardiovascular events in the last six months
* acute or chronic diseases limiting the capacity to understand and to participate in the trial
* masked hypertension
* white-coat hypertension
* secondary hypertension
* pregnancy
* breastfeeding
* concurrent participation in another trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-04; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Delta values for 24h ABPM between baseline and final ABPM measurements | 60 days

SECONDARY OUTCOMES:
Hypertension control | 60 days
Average of systolic and diastolic blood pressure at the end of the study. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C. Fuchs, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Fuchs SC, Ferreira-da-Silva AL, Moreira LB, Neyeloff JL, Fuchs FC, Gus M, Wiehe M, Fuchs FD. Efficacy of isolated home blood pressure monitoring for blood pressure control: randomized controlled trial with ambulatory blood pressure monitoring - MONITOR study. J Hypertens. 2012 Jan;30(1):75-80. doi: 10.1097/HJH.0b013e32834e5a4f. PMID 22134392